CLINICAL TRIAL: NCT04837092
Title: A Phase I/II Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of FR104, a Novel Antagonist Pegylated Anti-CD28 Fab' Antibody Fragment in de Novo Renal Transplant Patients
Brief Title: Phase I/II Study of FR104 First Administration In Patient With Renal Transplantation: FIRsT Study
Acronym: FIRsT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0007
Record Dates: First submitted 2020-12-03; First posted 2021-04-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplantation
Keywords: FR104; Renal transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FR104 Treatment (Experimental)
  Interventions: Drug: FR104

INTERVENTIONS:
Drug: FR104 — FR104 treatment administration at day 0, day 14 then every 28 days until month 12

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics (PK) of FR104 as well as its potential clinical effect on acute rejection prophylaxis and renal function in a de novo renal transplant population receiving an allograft from standard criteria donors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old
2. Signed and dated written informed consent prior to any study procedure
3. First kidney transplantation
4. Willing and able to participate to the study
5. Women of childbearing potential must use appropriate method(s) of contraception during the clinical trial (oral contraception, implant or intrauterine device) throughout the study period and for 90 days after the last dose of FR104
6. Women of childbearing potential must have a negative urinary pregnancy test the day of transplantation
7. All sexually active male subjects must agree to use an adequate method of contraception throughout the study period and for 90 days after the last dose of study drug and agree to no sperm donation until the end of the study, or for 90 days after the last dose of FR104, whichever is longer
8. Recipient of a kidney from deceased donor -
9. Recipient of a de novo kidney transplant able to start the immunosuppressive regimen at the protocol-specified time point
10. Recipients of a kidney with a cold ischemia time < 36 hours
11. Patients with French social security

Exclusion Criteria:

1. Recipient of a kidney from living donor
2. Patient at high immunological risk of rejection as determined for assessment of anti-donor reactivity:

   High TGI >20% or Presence of pre-formed DSA with MFI>500 (results 12 weeks prior to enrollment are acceptable if no blood transfusion or abortion occurred during this period)
3. Any retransplantation and combined transplantations
4. ABO incompatible transplantation
5. HIV-positive, EBV-negative or suffering active viral hepatitis B (AgHbs positive excluded) or hepatitis C, syphilis serology- positive recipient
6. CMV negative recipients of CMV positive donors (R-D+)
7. Patient with known history of tuberculosis
8. Uncontrolled concomitant infection or any other unstable medical condition (heart failure, severe liver disease, psychiatric disorders, substance abuse) that could interfere with the study objectives
9. A known allergy, hypersensitivity, or intolerance to the study drug, or to any of its components
10. Previous history of cancer (except appropriately treated non-melanoma skin cancer or localized cervical cancer, or other local tumors considered cured)
11. Pregnant woman or likely to become pregnant or nursing
12. Patient under guardianship or trusteeship
13. Patient participating in another interventional clinical trial
14. Live viral or bacterial vaccines/treatment agents given from 3 months prior to FR104 administration (12 months for BCG vaccine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Safety of FR104 - Adverse Events with a focus on infectious complications. In particular | Until Month 12
  Type, severity (grades 3 and 4 adverse effects)., number and percent of Adverse Events with a focus on infectious complications. In particular, the following cumulative incidences will be calculated: Incidence of bacterial, fungal, viral, or parasitic infection, incidence of new malignancies, lymphopenia, anemia, leucopenia, cytopenia or biochemical disturbances related to the study drug.

SECONDARY OUTCOMES:
Efficacy on Renal function | Month 6 and Month 12
  Calculated glomerular filtration rate (CKD EPI) at each visit.
Efficacy on Biopsy-proven acute rejection (BPAR) | Month 12
  Acute cellular rejection seen on renal biopsy for cause up to Month 12 (per Banff criteria 2017)
Efficacy on clinically-treated acute rejections | Month 12
  Graft acute rejection up to Month 12. Number of AE related to treatment. Incidence and grade of rejection proven on Biopsy analysed after M12.
Efficacy on steroid-resistant episodes | Month 12
  Steroid resistant episodes up to Month 12. Corticoresistant rejection up to month 12 defined as non response at day 5-6 after steroid boluses.
Efficacy on multiples rejection episodes | Month 12
  Rejection episodes up to Month 12. Number of rejection after M12. According to histology. Incidence of biopsy-proven rejection (by banff grade).
Efficacy on chronic allograft nephropathy | Month 12
  Chronic allograft nephropathy seen on renal biopsy for cause up to Month 12
Efficacy on graft survival | Month 12
  Renal dialysis or new kidney transplant up to Month 12
Treatment failure time | Month 12
  Time to treatment failure up to M12 (Biopsy-proven acute rejection, Graft Loss or Death)
Evaluate the first Biopsy-proven acute rejection time | Month 12
  Time to the first Biopsy-proven acute rejection
Evaluate the appearance of Donor specific Antibodies | Month 12
  Appearance of Donor specific Antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Blancho, Nantes, France